CLINICAL TRIAL: NCT02743052
Title: Optimal Anticoagulation Strategy In Stroke Related to CANCER (OASIS-CANCER Study)
Brief Title: Anticoagulation in Cancer Related Stroke
Acronym: OASIS-CANCER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SMC 2016-02-104
Record Dates: First submitted 2016-03-10; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-03

CONDITIONS: Cancer; Stroke
MeSH Terms: conditions — Neoplasms; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anticoagulation treatment. — Details of anticoagulation treatment information will be gathered including low molecular-weight heparin (enoxaparin 1 mg/kg) vs. NOAC (rivaroxaban 15 or 20 mg), vs. warfarin (target INR2.0-3.0) or no use of anticoagulation per physicians' decision and patients' conditions.

SUMMARY:
Purpose: Cancer associated intravascular coagulopathy is the primary mechanism of cancer-related stroke, particularly in those without conventional stroke etiologies. Randomized clinical trials have investigated efficacy of vitamin K-dependent oral anticoagulant (warfarin), low-molecular-weight heparin (LMWH) and non-vitamin K-dependent oral anticoagulant (NOAC) for the prevention of systematic venous thromboembolism. However, relatively little is known about the biological changes underlying intravascular coagulopathy and mechanisms of anticoagulation therapy in patients with cancer-related stroke. The aim of this study is to evaluate to determine the biological markers for intravascular coagulopathy causing stroke and for monitoring the effects of anticoagulation therapy, in patients with active cancer and stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years and older
* Acute ischemic stroke presented within 7 days of symptom onset
* Cancer related stroke: active cancer (diagnosis of cancer within 6 months of stroke onset, any treatment for cancer within the previous 6 months, or recurrent or metastatic cancer) and ischemic stroke which could not be explained by conventional stroke mechanisms including large artery atherosclerosis, cardioembolism, lacunar infarction, or other etiologies (e.g., dissection)
* Signed informed consent or appropriate signed deferral of consent where approved

Exclusion Criteria:

* Primary intracranial malignancy
* Incomplete workup for stroke etiology (either vascular or cardiologic studies)
* Any signs of infectious or immunological diseases which may influence plasma D-dimer levels
* Patients with stroke suspected to be caused by the tumor itself (i.e., tumor emboli) or cancer treatment (i.e., chemotherapy-induced stroke)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients with active cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Recurrent stroke or systemic embolism | up to 6 months
  Recurrent stroke (development of neurologic deterioration or a new symptom/sign and relevant new cerebral lesions documented by a neuroimaging study) or systemic embolism (objectively documented, symptomatic, recurrent deep-vein thrombosis, pulmonary embolism, or both ).

SECONDARY OUTCOMES:
90-days modified Rankin Scale score | examined at 90 days after stroke symptom onset in each patients
Effect of anticoagulation treatment | up to 14 days
  Effect of anticoagulation will be measured with D-dimer level during admission
Symptomatic hemorrhagic transformation | up to 6 months
  Symptomatic hemorrhagic transformation (newly developed cerebral hemorrhages that were temporally related to neurologic deterioration) or major bleeding up to 6 months (as defined by the International Society on Thrombosis and Haemostasis, J Thromb Haemost 2005;3:692-4)

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Bang, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No